CLINICAL TRIAL: NCT04772664
Title: Pilot-study: Probiotics and the Gut Brain Axis- Do Probiotics Interact With the Vagal Nerve? ProBIO-HRV-study
Brief Title: Probiotics and the Gut Brain Axis- Do Probiotics Interact With the Vagal Nerve?
Acronym: ProBIO-HRV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Allergosan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EK1019/2021
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Depressive Disorder, Major
Keywords: depression; vagal function; multispecies probiotic; heart rate variability
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants with Major Depression receiving a multi-strain probiotic (Experimental): Participants with Major Depression receiving a multi-strain probiotic
  Interventions: Dietary Supplement: Multispecies-Probiotic
- Participants mit Major Depression receiving a placebo (Placebo Comparator): Participants mit Major Depression receiving a placebo
  Interventions: Dietary Supplement: Placebo Supplement
- Healthy volunteers receiving a multi-strain probiotic (Experimental): Healthy volunteers receiving a multi-strain probiotic
  Interventions: Dietary Supplement: Multispecies-Probiotic
- Healthy volunteers receiving a placebo (Placebo Comparator): Healthy volunteers receiving a placebo
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Multispecies-Probiotic — Participants in intervention group receive 2x3g of a multistrain probiotic containing Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Bifidobacterium lactis W52, Lactobacillus acidophilus W22, Lactobacillus casei W56, Lactobacillus paracasei W20, Lactobacillus plantarum W62, Lactobacillus salivarius W24, Lactococcus lactis W19.
  Other Names: Omnibiotic-SR
  Arms: Healthy volunteers receiving a multi-strain probiotic; Participants with Major Depression receiving a multi-strain probiotic
Dietary Supplement: Placebo Supplement — Participants in the placebo group receive 2x3 gram of a placebo supplement not containing probiotic strains.
  Other Names: Placebo
  Arms: Healthy volunteers receiving a placebo; Participants mit Major Depression receiving a placebo

SUMMARY:
The purpose of this study is to investigate the effects of a multispecies probiotic on the function of the vagal nerve in patients with major depression and healthy participants in a single-center, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants giving written informed consent will be screened for eligibility for study entry and will be randomized in a double-blind manner to receive either a multistrain probiotic or a placebo for 3 months. At entry, 1 week after inclusion, 4 weeks after inclusion and 3 months (end of study) vagal activity will be measured using a 24hr electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* informed consenct
* confirmed diagnosis of depression according to ICD-10 or DSM-V
* age between 18 and 65 years

Exclusion Criteria:

* Suicidality
* no informed consent or no ability to provide consent
* cardiovascular disease
* pregnancy, breastfeeding
* alcohol or drug dependency
* other severe psychiatric or organic conditions (epilepsy, brain tumor, recent surgery)
* malignant diseases
* dementia (MMST<20)
* severe autoimmune-disorder or immunosuppression (systemic lupus, HIV, multiple sclerosis)
* antibiotic therapy in the last month
* misuse of laxative
* acute infections
* diarrhoea
* gastrointestinal surgeries (except appendectomy)
* no probiotic intake in the last 6 months
* no regular intake of other supplements, probiotics or antibiotics during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change of Vagal function | 4 measurements with 24-hr heart rate variability at study entry, one week after, 1 month after and after 3 months
  Heart rate variability parameters (logRSA; SDNN)

SECONDARY OUTCOMES:
Change of C-reactive protein (CRP) | 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  CRP is measured from serum samples with a Cobas analyzer.
Change of Interleukine-6 (IL-6) | 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  IL-6 is measured from serum samples with a Cobas analyzer.
Change of Oxytocin | 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  Oxytocin will be measured from serum samples using ELISA
Change of Gut microbiome analysis | 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  16S sequencing of gut microbiome samples, gut microbiota composition will be investigated with QIIME2 and characterized in terms of diversity (alpha-diversity, beta diversity) and differential bacterial abundance between time points.
Change of Body mass index | 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  Weight will be measured with a calibrated scale, height will be measured with a non expandable tape. BMI will be calculated using the formula [kg/m2].
Mini-international neuropsychiatric interview (M.I.N.I.) | at study entry
  short structured clinical interview which enables researchers to make diagnoses of psychiatric disorders according to DSM-IV or ICD-10
Change in Hamilton Scale for Depression (HAMD) | 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression
Beck Depression Inventory (BDI) | Change in 4 time points at study entry, one week after, 1 month after and 3 months (completion of the study)
  21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. The rating is as follows: 0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Change in Pittsburgh Sleep Quality Inventory (PSQI) | at study entry, after 7 days, after 4 weeks and after 3 months
  The PSQI is used to rate sleep quality. It includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Change in Adult Attachment Scale | at study entry, after 7 days, after 4 weeks and after 3 months
  The scale consists of 18 items scored on a 5 point likert-type scale. It measures adult attachment styles named "Secure", "Anxious" and "Avoidant", defined as:
  * Secure = high scores on Close and Depend subscales, low score on Anxiety subscale
  * Anxious = high score on Anxiety subscale, moderate scores on Close and Depend subscales
  * Avoidant = low scores on Close, Depend, and Anxiety subscales
Change in "Wiener Ernährungsprotokoll" | at study entry, after 7 days, after 4 weeks and after 3 months
  24-hr food recall
Change in International Physical Activity Questionnaire | at study entry, after 7 days, after 4 weeks and after 3 months
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients. There are no validated cut-offs.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No